CLINICAL TRIAL: NCT00224861
Title: Hypertension Telemanagement in African Americans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Dr. Joseph Finkelstein, Associate Professor of Medicine, Johns Hopkins University
Allocation: Randomized | Purpose: Treatment
Other Study IDs: 318; R01HL078579 (NIH)
Record Dates: First submitted 2005-09-21; First posted 2005-09-23 (Estimated); Last update posted 2013-03-25 (Estimated); Status verified 2013-03

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Self-Management

INTERVENTIONS:
Behavioral: Self-Management
Behavioral: Adherence

SUMMARY:
The specific goals of this project are to (1) refine the Home Automated Telemanagement (HAT) program according to the JNC 7 Report based on focus group review conducted by the key personnel, primary care providers, and patients and to fully implement the multidisciplinary model for hypertension telemanagement in African Americans as an adjunct of ambulatory care and (2) evaluate in a randomized clinical trial the impact of HAT on hypertension care delivery and on patients' clinical outcomes using both clinic- and patient-level variables. The comparison will be made with the standard of hypertension care recommended by the JNC 7 Report.

The following primary hypothesis related to clinic-level outcomes will be tested: Use of HAT will be associated (1) with improved proportion of treated patients who achieve blood pressure goals meeting JNC 7 recommendations, and (2) with a significant reduction in systolic and diastolic blood pressure. Researchers will also explore the impact of HAT on physician awareness and use of the hypertension treatment guidelines promulgated by the JNC 7 Report.

The following secondary exploratory hypothesis related to patient-level outcomes will be evaluated: The HAT program will have a positive impact on behavioral and cognitive factors that play an important role in the process of patient self-management, including hypertension treatment self-efficacy, health locus of control, health beliefs, and hypertension knowledge. Researchers will also investigate the impact of HAT on patients' compliance with multi-component treatment plans (including adherence to medication regimens and therapeutic lifestyle changes) and explore the effect of the HAT system on patients' ability to reach dietary, physical activity, weight control, and sodium consumption goals recommended by the JNC 7 Report.

During this study researchers will explore the impact of HAT on patient satisfaction with medical care, health-related quality of life, and health services utilization. Researchers will also assess acceptance of the HAT system by both patients and providers. Finally, researchers will perform a cost-effectiveness analysis of using the HAT system for hypertension control.

DETAILED DESCRIPTION:
BACKGROUND:

Recent studies demonstrated that successful chronic disease management requires a coordinated effort that includes health care providers who follow recent clinical guidelines in their everyday practice, educated patients who are adherent to their prescribed treatment plans, and comprehensive patient-provider communication. Studies employing telecommunication technologies have been successful in affecting the major components of chronic disease care, including physician practice patterns, patient adherence to therapy, and patient-provider communication. These studies were focused mainly on an improvement of a single component of the clinical care process. To date there have been no studies evaluating a coordinated approach that concurrently employs all of these components in an integrated framework linked to primary care. In this study researchers propose to evaluate a multi-component telemanagement system providing integrated support to both clinicians and patients in implementing hypertension treatment guidelines according to the JNC 7 Report.

DESIGN NARRATIVE:

Researchers will use the HAT system as a test platform for their intervention. The HAT system was developed to facilitate implementation of current clinical guidelines and to provide an integrated, multi-component chronic disease management intervention. HAT was designed as an Internet-based telemedicine system that (1) provides ongoing education to patients about their chronic disease, (2) helps patients follow their self-care plans, and (3) helps health care practitioners treat and monitor their patients' self-management process according to current clinical guidelines. The HAT system consists of (1) patient units (a computer or palmtop connected with a disease-specific testing device, such as a blood pressure monitor), (2) a HAT server that analyzes and stores self-testing results, and (3) clinician units that are used to review patient results on the Web. During each telecommunication session patients perform self-testing and receive structured disease-specific education, patient-tailored counseling, and advice on how to follow their individual self-care plans based on the current results of self-testing. The information for patients includes text, audio, and video components. In instances of patient noncompliance with self-testing, medication nonadherence, or failure to follow the physician-prescribed treatment plan, the system gives feedback to the patient to motivate better compliance and alerts the patient's physician and/or nurse who may contact the patient as well. This design can be easily adapted for any chronic condition by utilizing an appropriate disease-specific testing device and reprogramming decision support logic according to the particular disease management guidelines. In previous studies researchers have demonstrated (1) a high level of acceptance of the HAT system by patients from a low-income, inner-city area without previous computer experience, (2) acceptance of the system by physicians and nurses taking care of their patients, and (3) the validity of self-testing results in adult patients who used HAT. The system is currently being used to evaluate efficacy of home telemanagement of patients with asthma in the NIH- and ALA-funded studies. In this proposed study, researchers seek to advance their understanding of the applicability and utility of the HAT technology by focusing on its impact on African Americans with hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have a primary care provider at one of the clinics participating in the study
* Physician diagnosis of hypertension
* 21 years of age or older at the time of randomization
* African American by self-report
* Taking at least one medication prescribed for hypertension
* Poorly controlled blood pressure
* Understand spoken English
* Have a home telephone
* No other member of the household enrolled in the study

Exclusion Criteria:

* An identified secondary cause of hypertension
* Symptomatic myocardial infarction or stroke within the past 6 months
* Congestive heart failure (NYHA class III or greater)
* Significant renal impairment
* Diseases likely to lead to noncardiovascular death over the course of the study
* Evidence that the patient may move from the study area before the completion of the study
* Presence of any health condition that would preclude participation (e.g., psychiatric diagnosis or physical disability)
* Active drug use

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-09; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Finkelstein, Principal Investigator — University of Maryland